CLINICAL TRIAL: NCT06143930
Title: (Effect of Blood Flow Restriction Training on Muscle Strength and Gait Performance in Multiple Sclerosis Patients).
Brief Title: Blood Flow Restriction Training in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Habiba Zienhom Soubhy Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BFR in MS
Record Dates: First submitted 2023-10-25; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: MS

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (A) will receive therapeutic strengthening training program for lower extremities. (Active Comparator): low intensity strengthening exercise program
  Interventions: Other: strengthening ex
- The study group (B) will receive strengthening training with blood flow restriction (Active Comparator): the same selected low intensity resisted exercise program as group (A) with blood flow restriction
  Interventions: Other: strengthening ex with BFR training

INTERVENTIONS:
Other: strengthening ex with BFR training — Therapeutic strengthening training with blood flow restriction of trained limb.
  Arms: The study group (B) will receive strengthening training with blood flow restriction
Other: strengthening ex — Therapeutic strengthening training program for lower extremities.
  Arms: The control group (A) will receive therapeutic strengthening training program for lower extremities.

SUMMARY:
Traditional physical therapy resisted training for people with MS have been shown to be beneﬁcial; however, their usefulness has been limited by fatigue. The effect of blood flow restriction on strength and other measures of physical function was demonstrated in healthy populations and those with chronic disease. This study may add missing information to the existing literature and suggests directions for research on the effectiveness of BFR training on individuals with relapsing and remitting MS.

DETAILED DESCRIPTION:
Multiple sclerosis patients are characterized by impaired functional capacity which is related to reduce muscle strength affecting predominantly the lower extremity.

Resistance training (RT) has proven to be one of the interventions in MS patients showing a consistent and positive effect on muscle strength and on parameters directly related to lower extremity physical function (eg, walking performance and stair negotiation).

Training with blood flow restriction (BFR), is an increasingly common clinical intervention among physical therapists over the past decade and consistent with the evidence. It has been investigated in people with neurological disorders including stroke and incomplete Spinal Cord Injuries. Research is limited on the use of BFR for individuals with MS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were diagnosed with MS by a neurologist according to McDonald's criteria 2010
2. Expanded Disability Status Scale (EDSS) scores ranging from 2.5 to 5.5 .
3. Patient able to walk 100 meters or more.
4. No change within MS specific medication three months from the study.
5. Last Ms Attack from more than two months.

Exclusion Criteria:

1. Multiple sclerosis patients with other neurological or orthopedic problems.
2. Multiple sclerosis patients with systemic problems (cardiovascular or pulmonary diseases…).
3. Patients with cognitive impairment.
4. Pregnant female patients.
5. Patients in acute relapse stage.

   -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
muscle strength | one week after the end of treatment
  measure maximal torque production at a specified velocity of limb movement. measure torque of hip flexors , extensors , knee flexors and extensors

SECONDARY OUTCOMES:
gait performance by Two-dimensional (2D) Motion Analysis system | one week after the end of treatment
  kinematic analysis of gait (step length , stride length)

CONTACTS AND LOCATIONS:
Overall Officials: Habiba Zienhom, Principal Investigator — Cairo University; Dr.Moshera Hassan Darwish, professor, Study Director — professor of physical therapy,aculty of Physical therapy ,Cairo university; Dr Mohamed Soliman Al-Tamawy, professor, Study Director — professor of Neurology, Faculty of Medicine,Cairo university
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No